CLINICAL TRIAL: NCT01043250
Title: Effects of Atypical Antipsychotics on Appetite and Eating Behavior of Schizophrenia Patients: Analysis for Three Drugs, Olanzapine, Risperidone, and Aripiprazole, Known to Induce Different Degrees of Weight Gain
Brief Title: Effects of Atypical Antipsychotics on Appetite and Eating Behavior of Schizophrenia Patients
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Collaborators: Ministry of Health & Welfare, Korea (Other Government); Korea Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Kyung Sue Hong, M.D., Professor, Samsung Medical Center
Other Study IDs: 2009-04-005
Record Dates: First submitted 2010-01-04; First posted 2010-01-06 (Estimated); Last update posted 2011-07-25 (Estimated); Status verified 2011-07

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: schizophrenia; atypical antipsychotics; appetite; eating behavior
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Feeding Behavior

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Risperidone: Receiving risperidone treatment
- Olanzapine: Receiving olanzapine treatment
- Aripiprazole: Receiving aripiprazole

SUMMARY:
In this study, we are going to investigate quantitative and qualitative natures of appetite and eating-behavior changes induced by atypical antipsychotics, i.e., risperidone, olanzapine and aripiprazole, in schizophrenia patients.

DETAILED DESCRIPTION:
This is an observational study. 2 Self-report questionnaires assessing changes of appetite and eating behaviors after medication are applied to patients who have been receiving one of the three atypical antipsychotics. We are going to compare changes of appetite and eating behaviors after medication between three atypical antipsychotics and investigate the association between changes of appetite and eating behaviors and changes of weight after medication.

ELIGIBILITY:
Inclusion Criteria:

1. Patients meeting the DSM-IV criteria of schizophrenia, schizophreniform disorder, or schizoaffective disorder
2. Male and female patients aged 19~59
3. Patients receiving monotherapy with one of the three AAPs, i.e., olanzapine, risperidone, and aripiprazole for more than two and less than 24 months
4. Patients who had at least one-week antipsychotics-free periods before starting the above antipsychotics
5. Clinically stable and able to complete the questionnaires
6. Patients who sufficiently understand the objective of the study and sign informed consent form

Exclusion Criteria:

1. Patients having any medical illness or taking any medicine affecting appetite and body weight
2. Patients with severe and unstable medical, neurological or systemic illnesses
3. Patients having any comorbid psychiatric disorders including substance use disorders and eating disorders.
4. Pregnant or breast-feeding women

Ages: 19 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: outpatients clinic for schizophrenia
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2009-05; Primary Completion 2010-04 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Changes in appetite and eating behavior Rating Scales: Drug-related eating behavior questionnaire & Korean version of General Food Craving Questionnaire | between 2 and 24months after starting medication

SECONDARY OUTCOMES:
Body mass index (BMI) | between 2 and 24 months after starting medication

CONTACTS AND LOCATIONS:
Overall Officials: Kyung Sue Hong, MD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Background] Basson BR, Kinon BJ, Taylor CC, Szymanski KA, Gilmore JA, Tollefson GD. Factors influencing acute weight change in patients with schizophrenia treated with olanzapine, haloperidol, or risperidone. J Clin Psychiatry. 2001 Apr;62(4):231-8. doi: 10.4088/jcp.v62n0404. PMID 11379836